CLINICAL TRIAL: NCT06202105
Title: Comparison of Laparoscopic Versus Open Total Gastrectomy for Locally Advanced Gastric Cancer: a Prospective Randomized Control Trial
Brief Title: Comparison of Laparoscopic and Open Total Gastrectomy for Locally Advanced Gastric Cancer
Acronym: LOTA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Ho Chi Minh City (UMC) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LOTA
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic total gastrectomy (Experimental): 5 trocars were used. The gastrocolic ligament was divided along the border of the transverse colon. ligating the left gastroepiploic vessels to remove group 4sb.
  The right gastroepiploic vein was divided and right gastroepiploic and inferior pyloric artery were transected at their origin from the gastroduodenal artery to dissect group 6.
  The dissection was continued along the hepatoduodenal ligament to removed group 5 and group 12a and along the common hepatic artery to remove group 8a and along the celiac axis to remove group 9.
  The left gastric vein was divided and then the left gastric artery was vascularized to remove group 7.
  The dissection was continued upward along the splenic artery and its branches to remove group 11p,d and/or along the splenic hilum to remove group 10.
  The dissection was then conducted the right and left of the esophago-gastric junction to remove group 1,2.
  As a general rule, Roux en Y method was used for esophagoo-jejunal reconstruction for all cases
  Interventions: Procedure: Laparoscopic gastrectomy
- Open total gastrectomy (Active Comparator): An incision of 15~20 cm length is made in the abdominal midline . Standard total gastrectomy and omentectomy will be performed with D2 lymph node dissection (around common hepatic artery, celiac artery, along splenic artery, proper hepatic artery, and/or the splenic hilum) . Roux-en Y esophagojejunal anastomosis is performed for reconstruction.
  Interventions: Procedure: Laparoscopic gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic gastrectomy — Gastrectomy with laparoscopic approach

SUMMARY:
Evidence of implementation of laparoscopic total gastrectomy (LTG) for locally advanced gastric cancer (GC) remains inadequate. This study aimed to compare short- and mid-term outcomes of LTG versus open total gastrectomy (OTG) for cT2-4a GC.

DETAILED DESCRIPTION:
Gastric cancer (GC) is a significant public health issue worldwide. Surgical resection and lymphadenectomy is the first option for curative treatment of this disease. For tumors located in the middle and/or upper third of the stomach, open total gastrectomy (OTG) has long been the standard surgery.

While the advantage of laparoscopic distal gastrectomy over open distal gastrectomy for not only early gastric cancer (EGC) but also locally advanced gastric cancer (AGC) had been proven, the use of laparoscopic total gastrectomy (LTG) for GC, particularly for AGC, has not been widely accepted due to technical challenges with lymphadenectomy at the distal pancreas and the splenic hilum as well as the complexity of the esophago-jejunal reconstruction. Recently, there has been advancement in laparoscopic techniques and improved surgical experience, a standard procedure of LTG has been established, leading to increase utilization of LTG, especially for EGC. Two large RCTs, KLASS-03 in Korea and CLASS-02 in China, provided good evidence for the advantages of LTG for EGC. However, for AGC, some prior studies have demonstrated the safety of LTG compared to OTG but lacked significant data for survival. Until now, there have been no completed RCTs to determine the short- and long-term outcomes of LTG for AGC.

In the research center, LTG has been accepted as a standard procedure for EGC since 2008 and for AGC since 2013. In Vietnam and other low-to-middle-income countries, most GC was diagnosed in an advanced stage. It is needed to have evidence of the feasibility, safety, and oncological results of LTG for locally advanced GC. Investigators performed this study to compare the technical feasibility, short- and long-term outcomes of LTG versus OTG for stage T2-4a GC.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic finding by gastric endoscopy: confirmed gastric adenocarcinoma
* Age: 18 - 80 year old
* Tumor required total gastrectomy for radical treatment
* Preoperative cancer stage (CT scan stage): cT2-4aNanyM0
* ASA score: ≤ 3
* Informed consent patients (explanation about our clinical trials is provided to the patients or patrons, if patient is not available)

Exclusion Criteria:

* Concurrent cancer or patient who was treated due to other cancer before the patient was diagnosed gastric cancer
* Bulky lymph node andd/or Para-aortic lymph node metastasis
* Combined esophagectomy due to invading to the esophagus
* Pregnant patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2032-08-02 (Estimated); Study Completion 2032-08-02 (Estimated)

PRIMARY OUTCOMES:
3 year overall survival by Kaplan Mayer | 3 year after surgery
  The percentage of people in this study who are alive three years after surgery
3 year relapse-free survival by Kaplan Mayer | 3 year after surgery
  The percentage of people in this study who are alive without recurrence three years after surgery.

SECONDARY OUTCOMES:
operative morbidity | 30 days after surgery
  The rate of postoperative bleeding and the rate of postoperative leakage
operative mortality | 30 days after surgery
  The rate of postoperative dead
operative time | intraoperative
  The duration of a surgical procedure in minutes.
Resected lymph nodes | intraoperative
  The number of lymph nodes harvested after surgery
hospital stay | 30 days after surgery
  The number of days between surgery and discharge

CONTACTS AND LOCATIONS:
Locations (3):
- Vietnam (3):
  - Dong Nai General Hospital, Biên Hòa, Dong Nai
  - 108 Military Central Hospital, Hà Nội
  - University Medical Center Ho Chi Minh City, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Undecided